CLINICAL TRIAL: NCT05860140
Title: Prevention and Treatment of Malnutrition Among Home-living Older Adults Over 65 Years.
Brief Title: Preventing Malnutrition Among Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nord University (Other)
Responsible Party: Principal Investigator, Monica Christin Hansen, Principal Investigator, Nord University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 366924
Record Dates: First submitted 2023-04-17; First posted 2023-05-16 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-06

CONDITIONS: Malnutrition
Keywords: older adults; Disease-related malnutrition; Educational video
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): will get access to a six-minute educational video five days after being discharged from the hospital. The video is focusing on protein and energy meals for older adults.
  Interventions: Other: Education video
- Control group (No Intervention): Control group, not given any intervention

INTERVENTIONS:
Other: Education video — Six minutes long education video focusing on protein and energy meals
  Arms: Intervention group

SUMMARY:
This project aims to explore whether access to a digital education video can improve the nutritional situation of home-living older adults after being discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic and surgical in bedded patient patients in a selected regional hospital in Norway.
* Over 65 years old. Have their home address in one of nine selected municipalities in Nordland county.
* home living and due to return home after discharge directly from the hospital or after a short-term training stay at a training centre before returning home.
* Could read and understand Norwegian.
* Have consent competence.
* Have a Body mass index less than 24.

Exclusion Criteria:

* Patients patients only receiving liquid diet such as tube feeding
* terminal-ill patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life Using Rand 36 Questionnaire | Change in Health related quality of life Using Rand 36 Questionnaire after 3 months
  Using Rand 36 Questionnaire

SECONDARY OUTCOMES:
Body fat | Change in Body mass index after 3 months
  Body fat will be measured by Body mass index (BMI). weight (in kg) and height (in cm) will be combined to report BMI in kg/m^2.
Readmissions to hospital after discharge from the hospital | Registration of Readmissions 3 months after
  Readmissions after discharge from the hospital will be meassured three months after discharge
Muscle Strength | Change in Hand Grip Strength (muscle strenght) after 3 months
  Measure Muscle Strength in kg using Saehan Hydraulic Hand Dynometer for Hand Grip strength in both hands.
The mid-arm circumference | Change in The mid-arm circumference after 3 months
  The mid-arm circumference (MAC) will be measured in cm with a measuring tape. This will be done of the left upper arm measured at the midpoint between the tip of the shoulder and the tip of the elbow
Subcutaneous fat | Change in Subcutaneous fat after 3 months
  Subcutaneous fat will be measured by Triceps skinfold thickness (TFS). This will be done by a in millimetres with a VirtuFits Digital Fat Caliper skinfold in the triceps of the left arm.
Muscle protein mass | Change in Muscle protein mass after 3 months
  Muscle protein mass will be measured by the mean arm muscle circumference (MAMC) calculated according to the formula: MAMC (cm) = MAC (cm) - (3,14 X TFS x 0,1)

CONTACTS AND LOCATIONS:
Locations (1):
- Monica Christin Hansen, Bodø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen MC, Uhrenfeldt L, Ingstad K, Pedersen PU. The feasibility of an education video for preventing disease-related malnutrition among home-living older adults after discharge from a surgical hospital department - a randomised controlled feasibility trial. Pilot Feasibility Stud. 2025 Dec 5;12(1):6. doi: 10.1186/s40814-025-01745-y. PMID 41351135
- [Derived] Hansen MC, Ingstad K, Uhrenfeldt L, Pedersen PU. Assessing the impact of a nutrition educational video on health-related quality of life in older home-living adults after discharge from a surgical hospital department: a randomised controlled pilot trial. BMC Nutr. 2025 Nov 25;11(1):230. doi: 10.1186/s40795-025-01203-1. PMID 41291959